CLINICAL TRIAL: NCT00214864
Title: A Pilot Study of Taxotere (Docetaxel) Combined With Xeloda (Capecitabine) in the Treatment of Metastatic Breast Cancer
Brief Title: A Study of Weekly Taxotere and Xeloda in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research Network (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRN-003
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Taxotere (docetaxel); Xeloda (capecitabine)
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel, capecitabine — cohort 1 = capecitabine 900mg/m2 BID POx14 days and docetaxel 36mg/m2 day1&8 cohort 2 = capecitabine 650mg/m2 BID POx14 days and docetaxel 30mg/m2 day1&8 cohort 3 = capecitabine 850mg/m2 BID POx14 days and docetaxel 30mg/m2 day1&8

SUMMARY:
The purpose of this study is to attempt to find better tolerated doses and schedules of this highly effective combination chemotherapy regimen.

DETAILED DESCRIPTION:
Combination chemotherapy has advantages over monochemotherapy due to the higher response rates that can often be obtained; by using agents with non-overlapping toxicity profiles, these responses can be achieved with less toxicity than maximally tolerated doses of single agents. One significant advantage of capecitabine/weekly docetaxel combination chemotherapy is that both agents appear to have a toxicity profile appropriate for palliative therapy of advanced breast cancer. This trial will utilize the usual schedule of capecitabine used in the USA, which is two times per day oral dosing for 14 days but at a reduced dose in hopes of decreasing toxicities. Docetaxel will be given weekly at a dose of 35 mg/m2 X 2 with a one-week rest to coincide with the 14-day schedule of capecitabine.

The primary objective is to evaluate the overall response rate (complete and partial responses) according to the RECIST criteria of the combination of capecitabine and docetaxel with the selected schedule in patients with advanced and/or metastatic breast cancer. The secondary objectives are to evaluate tolerability, time to tumor progression, and time to treatment failure of the combination of capecitabine and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histopathologically proven metastatic breast cancer.
* Patients 18-75 years old
* Performance status: Karnofsky > 70%
* Patients must have measurable disease. Patients with only blastic bone lesions are ineligible.
* Adequate bone marrow, liver, renal and cardiac functions defined as:
* Ability to understand the study and give informed consent.
* Patients may not have received more than one prior chemotherapy for metastatic breast cancer. 5-FU or Taxol given as part of an adjuvant regimen will not render the patient ineligible.

Exclusion Criteria:

* Patients with brain metastasis, adequately treated and stable and not requiring continued steroid medication will be eligible if no progression for > 3 months.
* Patients who have received any anti-cancer investigational agent in the month prior to inclusion.
* Patients previously treated with docetaxel(Taxotere)or capecitabine (Xeloda).
* Patients with lack of physical integrity of the upper gastrointestinal tract, inability to swallow tablets or those who have malabsorption syndrome.
* Patients with renal impairment (creatinine clearance below 30 ml/min calculated according to Cockcroft and Gault, see Appendix D), since capecitabine is contraindicated in patients with severe renal impairment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-12; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To find the lowest tolerable efficacious dose of the docetaxel/capecitabine combination | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Vogel, MD, Principal Investigator — Cancer Research Network, Inc; Elizabeth Tan-Chiu, MD, Study Chair — Cancer Research Network, Inc.
Locations (1):
- Cancer Research Network, Inc., Plantation, Florida, United States